CLINICAL TRIAL: NCT02834156
Title: Impact Assessment of Positioning on Pain Sensitivity During a Lumbar Puncture in Children
Brief Title: Impact of Child Positioning on Pain During a Lumbar Puncture
Acronym: PHIPA-PEPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-PP-05
Record Dates: First submitted 2016-07-08; First posted 2016-07-15 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LP in a seated position then LP in a lying position (Other): Patients will have first a lumbar puncture (LP) in a seated position then a LP in a lying position
  Interventions: Other: LP in a seated position then LP in a lying position
- LP in a lying position then LP in a seated position (Other): Patients will have first a lumbar puncture (LP) in a lying position then a LP in a seated position
  Interventions: Other: LP in a lying position then LP in a seated position

INTERVENTIONS:
Other: LP in a seated position then LP in a lying position
  Arms: LP in a seated position then LP in a lying position
Other: LP in a lying position then LP in a seated position
  Arms: LP in a lying position then LP in a seated position

SUMMARY:
This protocol is a pilot study on standard care. The main goal is to assess the impact of positioning on lumbar puncture process especially on pain sensitivity in children.

It's a prospective, monocentric, randomized, open-label, cross-over study. Inclusion period is one year, and number of inclusions forecasted is about 30. Each patient will have one LP in a seated position and one in a lying position.

DETAILED DESCRIPTION:
In Pediatric Oncology Hematology, invasive procedures such lumbar punctures or myelograms are essential to diseases diagnosis and treatment.

In hematological malignancies, lumbar punctures are particularly frequent as the therapy processes. Despite a good analgesia, this repeated procedure can generate pain, anxiety, apprehension leading to an increasing difficulty in the procedure realization.

Two positions are possible to carry out lumbar puncture: seated or lying position.

The main goal of this study is to assess the impact of the child positioning during the lumbar puncture process in term of pain, anxiety and stress.

This study is a prospective, monocentric, randomized, open-label, cross-over study. Inclusion period is 1 year, 30 patients will be included from 2 to 18 years old.

Each patient will have 2 LP one in seated and one in lying position in a specific order determined by randomization.

All data regarding pain and anxiety will be collected the day of LP. Patients will be re contacted 48 hours and 15 days after LP procedure in order to evaluate complications such post-lumbar puncture syndrome or hematoma. The main analysis will be done on intent-to-treat-analysis basis and will compare pain intensity between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 18 years old
* Patients requiring at least 2 therapeutic lumbar punctures
* Patients able to receive analgesic procedure according to 20005 good practices recommendation
* Presence of one parent during LP procedure
* Child able to use assessment scales
* LP realized with a 20 G needle
* Platelets > 50000
* Child with prior clinical examination
* Affiliated to a health care insurance regimen

Exclusion Criteria:

* Seated or lying position impossible
* Lumbar puncture contraindication
* Patient or parent opposition to second LP realization in the required position
* Clotting trouble on LP day not allowing the LP procedure

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity during the lumbar puncture procedure. | duration of the procedure
  It will be evaluated throw specific pain assessment scales according to patient age

SECONDARY OUTCOMES:
Anxiety during the lumbar puncture procedure on a scale of one to ten | duration of the procedure
Time of the lumbar puncture procedure | duration of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No